CLINICAL TRIAL: NCT03585803
Title: A Dose Blocked-Randomized, Single-Blind, Placebo-Controlled and Dose-Escalation Phase I Clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetic/Pharmacodynamic Characteristics of KMRC011 After Intramuscular Administration in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetic/Pharmacodynamic Characteristics of KMRC011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intron Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMRC011-01
Record Dates: First submitted 2018-06-03; First posted 2018-07-13 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Acute Radiation Syndrome
MeSH Terms: conditions — Acute Radiation Syndrome | interventions — KMRC011; KPNA1 protein, human

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- KMRC011 5μg or Placebo (Other): Cohort 1
  Interventions: Drug: KMRC011 5μg or Placebo
- KMRC011 10μg or Placebo (Other): Cohort 2
  Interventions: Drug: KMRC011 10μg or Placebo
- KMRC011 15μg or Placebo (Other): Cohort 3
  Interventions: Drug: KMRC011 15μg or Placebo
- KMRC011 20μg or Placebo (Other): Cohort 4
  Interventions: Drug: KMRC011 20μg or Placebo
- KMRC011 25μg or Placebo (Other): Cohort 5
  Interventions: Drug: KMRC011 25μg or Placebo

INTERVENTIONS:
Drug: KMRC011 5μg or Placebo — Intramuscular Injection of KMRC011 5μg or Placebo(Normal Saline) 0.1ml
  Other Names: Cohort 1
  Arms: KMRC011 5μg or Placebo
Drug: KMRC011 10μg or Placebo — Intramuscular Injection of KMRC011 10μg or Placebo(Normal Saline) 0.2ml
  Other Names: Cohort 2
  Arms: KMRC011 10μg or Placebo
Drug: KMRC011 15μg or Placebo — Intramuscular Injection of KMRC011 15μg or Placebo(Normal Saline) 0.3ml
  Other Names: Cohort 3
  Arms: KMRC011 15μg or Placebo
Drug: KMRC011 20μg or Placebo — Intramuscular Injection of KMRC011 30μg or Placebo(Normal Saline) 0.4ml
  Other Names: Cohort 4
  Arms: KMRC011 20μg or Placebo
Drug: KMRC011 25μg or Placebo — Intramuscular Injection of KMRC011 45μg or Placebo(Normal Saline) 0.5ml
  Other Names: Cohort 5
  Arms: KMRC011 25μg or Placebo

SUMMARY:
This trial is designed to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic of KMRC011 injection in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A male whose age is between 19 and 55 years of age
* A person whose body mass index is between 18.5 and 27 kg/m2 at screening
* A person who has the ability and willingness to participate in the clinical trial
* A person who voluntarily agrees with the clinical trial after hearing and fully understanding the detailed explanation of this clinical trial

Exclusion Criteria:

* A person who has a clinically significant disease or history of liver, kidney, neuropsychiatry, immune system, respiratory system, endocrine system, hematology*oncology system, cardiovascular system, etc.(In the case of liver disease items, it includes subjects who have hepatitis virus)
* A person who has clinical history of hypersensitivity reactions to the major components or constituents of investigational product or other clinically significant hypersensitivity reactions to drugs or foods, or those with allergic diseases requiring treatment
* A person with infectious disease or severe trauma within 21 days of the randomization date
* A person whose serum AST, ALT or γ-GT levels exceed 1.5 times the upper limit of the reference range at screening
* A person whose QTcF on the electrocardiogram exceeds 430 msec or who has a clinically significant abnormal rhythm at screening
* A person with a glomerular filtration rate less than 60 mL/min/1.73 m2 calculated from serum creatinine at screening
* A person with a systolic blood pressure less than 100 mmHg, greater than 150 mmHg, diastolic blood pressure less than 60 mmHg, or greater than 100 mmHg at screening
* A person with thrombocytopenia or coagulopathy which should not be given intramuscular injection
* A person whose weekly average drinking amount exceeds 140g of alcohol per week
* A person whose daily average smoking amount exceeds 10 per day
* A person who have received a drug that can significantly affect the absorption, distribution, metabolism or excretion of the investigational product within 14 days of the injection
* A person who has the history of substance abuse or positive urine screening test
* A person who have received a investigational product or a bioequivalence study drug within at least 90 days prior to the randomization
* A person who donated whole blood within 60 days before the randomization, or donated components of blood within 30 days
* A person who dose not have a medically approved contraceptive during the trial and has a plan to provide sperm
* A person who has clinically significant abnormalities from clinical laboratory test
* A person who is deemed ineligible for clinical trials by the investigator

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse event or adverse drug reaction | Up to 7±1 days after injection
Number of subjects with clinically significant changes in hematology test result after injection | Up to 7±1 days after injection
Number of subjects with clinically significant changes in blood chemistry test result after injection | Up to 7±1 days after injection
Number of subjects with clinically significant changes in urinalysis test result after injection | Up to 7±1 days after injection
Number of subjects with clinically significant changes in blood coagulation test result after injection | Up to 7±1 days after injection
Number of subjects with clinically significant changes in ECG (Electrocardiogram) after injection | Up to 7±1 days after injection
Number of subjects with clinically significant changes in vital sign after injection | Up to 7±1 days after injection
Number of subjects with clinically significant physical abnormality after injection | Up to 7±1 days after injection
Maximum serum concentration (Cmax) of KMRC011 | Pre-dose(0 hours) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post-dose
Time of the maximum serum concentration (Tmax) of KMRC011 | Pre-dose(0 hours) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post-dose
Area under the serum concentration versus time curve, from time 0 to the last measurable concentration (AUC0-t) of KMRC011 | Pre-dose(0 hours) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post-dose
Area under the serum concentration versus time curve from time 0 to infinity (AUCinf) of KMRC011 | Pre-dose(0 hours) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post-dose
Percentage of AUCinf due to extrapolation from time of last measurable concentration to infinity (AUCextra) of KMRC011 | Pre-dose(0 hours) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post-dose
Apparent clearance (CL/F) of KMRC011 | Pre-dose(0 hours) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post-dose
Apparent volume of distribution (Vd/F) of KMRC011 | Pre-dose(0 hours) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post-dose
Terminal half-life (t1/2) of KMRC011 | Pre-dose(0 hours) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post-dose
Maximum effect over the time span specified (Emax) of G-CSF | Pre-dose(0 hours) and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48 hours post-dose
Maximum effect over the time span specified (Emax) of IL-6 | Pre-dose(0 hours) and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48 hours post-dose
Area under the effect versus time curve, from time 0 to the last measurable concentration (AUEC0-t) of G-CSF | Pre-dose(0 hours) and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48 hours post-dose
Area under the effect versus time curve, from time 0 to the last measurable concentration (AUEC0-t) of IL-6 | Pre-dose(0 hours) and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48 hours post-dose

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of KMRC011 | Until the study completion, approximately up to 35 weeks
  A dose that is one level lower than the dose which Dose Limiting Toxicity (DLT) incidence is 33% or more is determined as a Maximum Tolerated Dose (MTD). If the Dose Limiting Toxicity (DLT) incidence is lower than 33% at all doses level, we conclude Maximum Tolerated Dose (MTD) cannot be determined.

OTHER OUTCOMES:
Number of subjects who expressed Anti-Drug (KMRC011) Antibody (ADA) | Up to 28±2 days after injection

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Ryul Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Gangnam-gu, Seoul, South Korea